CLINICAL TRIAL: NCT05239169
Title: A Phase II Study of Immunotherapy With Durvalumab and Tremelimumab in Combination With Capecitabine or Without Capecitabine in Adjuvant Situation for Biliary Tract Cancer
Brief Title: Immunotherapy With Durva and Treme With or Without Capecitabine in Adjuvant Treatment for Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADJUBIL; AIO-HEP-0421/ass (Other: AIO)
Record Dates: First submitted 2021-12-20; First posted 2022-02-14 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer (CCA); Intrahepatic Cholangiocarcinoma; Hilar Cholangiocarcinoma; Distal Cholangiocarcinoma; Gall Bladder Carcinoma
Keywords: Biliary Tract Cancer; CCA
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Klatskin Tumor; Gallbladder Neoplasms | interventions — durvalumab; tremelimumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: Treatment consists of durvalumab and tremelimumab with or without capecitabine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Cape+Durva+Treme (Experimental): Capecitabine + Durvalumab + Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Capecitabine
- B: Durva+Treme (Active Comparator): Durvalumab + Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab at a fixed dose of 1500 mg as an IV infusion over 1 hour, on day 1 together with the Tremelimumab infusion. Durvalumab only infusion to be repeated every 4 weeks for a maximum of 12 months on day 1 of each cycle.
Drug: Tremelimumab — Tremelimumab at a fixed dose of 300 mg as an IV infusion over 1 hour on day 1 of cycle 1.
Drug: Capecitabine — Capecitabine at 1250 mg/m² p.o. twice a day on days 1 to 14 of a 3-weekly cycle (eight cycles).
  Arms: A: Cape+Durva+Treme

SUMMARY:
This is an interventional, prospective multicenter, open-label, phase II study in patients after curative surgery for BTC in a classic adjuvant situation, consisting of a two arm feasibility pilot part with a randomized pick-the-winner design and an option to proceed into a randomized phase 2/3 trial in order to compare the winner with the current SOC (capecitabine).

DETAILED DESCRIPTION:
The primary objective is to assess the anti-tumor activity of the combination of durvalumab and tremelimumab with or without capecitabine by the recurrence-free survival rate after 12 months (RFS@12).

Secondary objectives are to assess the efficacy by recurrence-free surviaval (RFS) and overall survival (OS); to assess safety of the combination treatments (AEs, impact on liver function, use of subsequent therapies); to assess quality of life (QoL).

Exploratory objective is to perform correlation analysis between selected molecular parameters and clinical data to identify molecular biomarkers predictive for RFS and OS.

Patients will be stratified according to the tumor site (ICC vs. ECC vs. gallbladder) and resection status (R0 vs. R1).

In this pilot trial phase, a pick the winner design is applied to determine wether treatment with durvalumab and tremelimumab in combination with or without capecitabine is more promising.

In the initial pilot phase, 40 patients with histologically proven and curatively resected biliary tract cancer (intrahepatic, hilar or distal CCA as well gallbladder carcinoma) without metastatic disease, will be enrolled in a 1:1 randomized design (i.e. 20 patients per Arm).

Patients will be recruited from up to 15 sites and patients withdrawn from the trial will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, including participation in optional translational research if applicable, and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Histologically proven and curatively resected biliary tract cancer (intrahepatic, hilar or distal CCA as well gallbladder carcinoma) without metastatic disease, in the adjuvant situation (R0/R1) up to 16 weeks from surgery.
3. Men or women* ≥ 18 years at time of study entry.

   *There is no data that indicates a specific gender distribution. Therefore, patients are included regardless of their gender.
4. Performance status (PS) ≤ 1 (ECOG scale),with no deterioration over the previous two weeks prior to baseline.
5. Must have a life expectancy of at least 12 weeks
6. Appropriate hematological, hepatic and renal function:

   * Absolute number of neutrophils (ANC) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL (5.58 mmol/L)
   * Total bilirubin ≤ 1.5 times the upper limit of normal (UNL) or ≤3 x ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia)
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL
   * Serum creatinine ≤ 1.5 x UNL or creatinine clearance (measured by 24h urine) ≥ 40 mL / min (i.e., if the serum creatinine level is > 1.5 x UNL, then a 24-h urine test must be performed to check the creatinine clearance to be determined).
7. Adequate coagulability, as determined by the International Normalized Ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 5 seconds above the UNL (unless anti-coagulation therapy has been given). Patients receiving warfarin / phenoprocoumon must be switched to low molecular weight heparin and before starting study-specific procedures.
8. Patients of reproductive age must be prepared to use a suitable contraceptive method during the study and up to 3 months after the end of treatment. A suitable method of contraception is defined as surgical sterilization (e.g., bilateral fallopian tube ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double barrier methods (each two-fold combination of intrauterine pessary, condom for men, or women with spermicidal gel, Diaphragm, contraceptive sponge, cervical cap). Women of child-bearing potential must have a negative serum pregnancy test within the last 7 days prior to the start of study therapy.

   Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving IMP and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational products (durvalumab and tremelimumab).

   Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception).
9. Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Presence of tumors other than biliary tract cancer or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. Patients who have received curative treatment for other tumors and have been disease-free for at least 5 years at the time of screening are eligible for enrollment.
2. Metastatic biliary tract cancer disease.
3. Simultaneous, ongoing systemic immunotherapy, chemotherapy, or hormone therapy not described in the study protocol.
4. Simultaneous treatment with a different anti-cancer therapy other than that provided for in the study (excluding palliative radiotherapy only for symptom control)
5. Previous therapy with a PD-1, PD-L1 inhibitor (including durvalumab) or CTLA4 inhibitor (including tremelimumab) or classical chemotherapy agents like platinum, fluoropyrimidine or gemcitabine based regimens.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the LKP.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the LKP.
7. Stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
8. Known allergic / hypersensitive reactions to at least one of the treatment components.
9. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent within the last 12 months prior to the start of the study.
11. Presence of an active, uncontrollable infection.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
13. Active disseminated intravascular coagulation.
14. Any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
15. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
16. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
17. History of active primary immunodeficiency
18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival at 12 months (RFS@12). | 12 months
  Recurrence free survival at 12 months (RFS@12) will be defined as the proportion of allocated subjects without any recurrence/progression and alive at 12 months after the date of treatment allocation.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | 30 months
  Recurrence-free survival (RFS) will be determined as time from the date of treatment allocation to the date of (1) any recurrence/progression (local or regional [including invasive ipsilateral tumor and invasive locoregional tumor], or distant) or (2) death due to any cause.
Overall survival (OS) | 30 months
  Overall survival (OS) will be determined as time from the date of treatment allocation to the date of death due to any cause. A subject who has not died will be censored at last known date alive.
Safety: (serious) adverse events | 30 months
  Safety assessments will include adverse events. All observed toxicities and side effects will be graded according to NCI CTCAE v5.0 for all patients and the degree of association of each with the study treatment assessed and summarized. Treatment related serious adverse events rate (SAE) will be determined.
QoL QLQ-C30 | 30 months
  QoL will be assessed by the EORTC QLQ-C30 questionnaire in itsmost current version.
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment.
  EORTC QLQ C30 (30 questions) regarding body fitness, daily routines, restrictions at work and hobby, appetite, fatigue, cough, breathlessness, pain, tiredness, body conditions, state of health and Quality of life.
QoL BIL21 | 30 months
  QoL will be assessed by the EORTC QLQ-BIL21 questionnaire in its most current version.
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment.
  EORTC QLQ BIL21 (21 questions) regarding eating habits, body fitness, fatigue, pain, tiredness and mental health.
QoL EQ-5D-5L | 30 months
  QoL will be assessed by the QoL EQ-5D-5L questionnaire in its most current version.
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment.
  EQ 5D-5L (6 questions) about mobility, sorrows, daily routine, pain, anxiety and health perception.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Thorsten O. Götze, Prof. Dr., Principal Investigator — Institut für Klinische Krebsforschung IKF GmbH
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.